CLINICAL TRIAL: NCT03032679
Title: Postoperative Pain Severity, Incidence Of Chronic Pain And Its Impact On Daily Function Following Total Knee Replacements (TKR) At A Tertiary Cancer Institute
Brief Title: Pain and Impact of Chronic Pain on Function After Total Knee Replacements
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Aparna Chatterjee, Professor, Tata Memorial Centre
Other Study IDs: 1780
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative; Pain, Chronic; Osteogenic Sarcoma; Knee Arthropathy
Keywords: pain, acute, chronic, knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Osteosarcoma; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group of patients: Non interventional study. Observational with questionnaires
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — No intervention

SUMMARY:
After Institutional Review Board approval, adult patients scheduled for total knee arthroplasty (TKA) will be enrolled into the study after obtaining informed consent over a 24 month period. Interim analyses of cases who have completed the 6 month follow up as on 31st October, 2017 will be analyzed as part of the co- principle investigator's thesis. All consenting patients will be assessed for pain preoperatively, the first 3 post-operative days, at 1, 4 and 6 months from the date of surgery. Pain scores will be assessed using the Numerical Rating Scale during the 3 postoperative days. Pain will be managed by the Acute Pain Service team as per standard protocols.

The Brief pain inventory (BPI) (short form with translations, obtained with permission from MD Anderson), which assesses pain severity and its impact on daily functions will be administered to the patient in a language familiar to them, preoperatively, at 1, 4 and 6 months postoperatively.

The Musculoskeletal Tumour Society Score (MSTS) which evaluates the functional condition (impairment) after completed tumour treatment will be estimated at the end of 6 months from the date of surgery The painDETECT questionnaire (PD-Q) a quick, simple and reliable screening tool to identify the likelihood of a neuropathic pain component in patients and validated in various languages including Hindi and Marathi will be administered preoperatively and at 1, 4 and 6 months after surgery.

Details of postoperative chemotherapy and radiation will also be obtained from patient's notes and the electronic medical record. If the patient cannot follow up at the said intervals, the pain scores would be obtained telephonically and the BPI and PD-Q forms in prepaid envelopes would be given to them at discharge which they would have to duly fill in and post them to the given address at the appropriate intervals if they cannot visit the pain clinic. At the 6th month of follow up, they would be requested to visit the pain clinic for an assessment of MSTS score and completing the BPI and PD-Q.

INCLUSION CRITERIA:-

* Adult patients above 18 years of age, undergoing TKR
* Literate: able to read and write in at least one of the following languages English, Hindi and Marathi
* Willing to fill forms and post them and/or answer questions on phone

EXCLUSION CRITERIA:-

* Refusal of consent
* Cognitively impaired
* Revision TKRs (including cases with wound wash and nail spacer cementing)

DETAILED DESCRIPTION:
INTRODUCTION:- A Total Knee Replacement (TKR) or arthroplasty (TKA) is a complex procedure that requires an Orthopedic Surgeon to make precise measurements and skillfully remove the diseased portions of the bone, in order to shape the remaining bone to accommodate the knee implant. Knee Replacement Surgery is most commonly performed in people with advanced osteoarthritis and should be considered when conservative treatments have been exhausted. Oncologic TKRs are different from the routine TKRs in a way that the former involves a wide local resection of the bone and soft tissues, ranging from 10 to 20 cm, resection of muscles like the head(s) of biceps femoris, the gastrocnemius muscle, the intermuscular septa, the joint capsule, etc. to ensure negative margins along with the complete resection of the tumour, followed by a reconstruction of almost the same length as that resected, to restore function.

The most common indication for doing oncologic TKR is Osteogenic Sarcoma (OGS) of and around the knee joint. The distal femur and proximal tibia are among the most common sites for primary bone tumor. OGS is the most common bone cancer in the world in children and adolescents, and the eighth-most common form of childhood cancer, accounting for 4% of all childhood cancers worldwide. In India, the incidence varies from 4.7% to 11.6%, where this malignancy is associated with significant morbidity and mortality. Additional treatment involves chemotherapy which further delays the healing and recovery of the patient.

Surgery is a known risk factor for development of Chronic Post Surgical Pain(CPSP) which as per the definition given by Macrae and Davies, is defined by

* Pain developing after a surgical procedure.
* Pain of at least 2 months' duration.
* Other causes of pain excluded (e.g.- malignancy, infection, etc.).
* Pain continuing from a pre-existing pain problem excluded.

CPSP is a well known risk factor in many surgeries like (but not exclusive of)-

* Mastectomy (Incidence of chronic pain = 11-57%)
* Amputation (30-85%)
* Inguinal hernia(5-63%)
* Cholecystectomy (3-50%)

CPSP develops after a surgical procedure or increases in intensity after the surgical procedure. Literature on TKR surgeries indicated for osteoarthritis, report that although many patients report a good outcome after their total knee replacement, at a time when recovery should have been achieved, about 10-34% of patients undergoing TKR for osteoarthritis report moderate to severe CPSP. In around 30% of patients with CPSP, the origin of CPSP might be neuropathic. Neuropathic pain is more severe and adversely affects the quality of life of patients. TKR on its own may cause neuropathic pain postoperatively due to local nerve damage, often to the infrapatellar branch of the saphenous nerve or due to local inflammation. Risk factors associated with the operation include increased duration of surgery and tourniquet time, revision surgery, TKA versus unicompartmental arthroplasty and intraoperative nerve damage. Oncologic TKRs are more extensive and include much morbid excisions, and consequently may be presumed to have a similar if not a greater incidence of CPSP. Some of the risk factors for CPSP include the following (but not exclusive of)-

* Pain, moderate to severe, lasting more than 1 month
* Repeat surgery
* Younger age (adults)
* Surgical approach with risk of nerve damage
* Neurotoxic chemotherapy

Preoperative pain is consistently found to be a predictor for persistent postsurgical pain, which might reflect an independent risk factor but could well be a manifestation of predisposing factors.

Tata Memorial Hospital, a tertiary cancer institute is a 629 bedded hospital and conducts approximately 6000 surgeries per year out of which approximately 100 TKRs are performed per year. Analgesia peri-operatively is provided by an epidural infusion of a combination of local anaesthetic and an opioid or intravenous opioids with non-steroidal anti-inflammatory analgesics and paracetamol as appropriate. Postoperatively, if inserted, epidural analgesia is continued for up to 3-4 days to help mobilization & physiotherapy. In the absence of an epidural, around the clock analgesics with or without an opioid administered by means of an Intravenous Patient Controlled Analgesia (IVPCA) device is instituted. These patients are visited by the acute pain service team to address pain issues for the first 3 postoperative days or sometimes longer.

STUDY DESIGN:- Prospective and Observational study

METHODS and MATERIALS:- After Institutional Review Board approval, adult patients scheduled for TKR surgeries will be enrolled into the study after obtaining their informed consent over a 24 month period. However, interim analyses of all cases who have completed the 6 month follow up as on 31st October, 2017 would be analyzed as part of the co- principle investigator's thesis. All consenting patients will be assessed for their pain preoperatively and for the first 3 post-operative days, and at 1, 4 and 6 months from the date of surgery. Pain scores will be assessed using the Numerical Rating Scale during the 3 days after surgery. Pain will be managed by the Acute Pain Service team as per the standard management protocols.

The Brief pain inventory (BPI), (short form with translations, obtained with permission from MD Anderson), which assesses the severity of pain and the impact of pain on daily functions will be administered to the patient in the language familiar to them, preoperatively, at 1, 4 and 6 months postoperatively. The BPI is a useful instrument to assess the severity of pain and impact of pain on daily functions in patients with pain from chronic diseases, conditions such as cancer, osteoarthritis and low back pain, or with pain from acute conditions such as postoperative pain. The short form comprises of nine questions related to the severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. It has been widely used and validated in several languages the world over.

The Musculoskeletal Tumour Society Score (MSTS) evaluates the functional condition (impairment) after completed tumour treatment will be estimated at the end of 6 months from the date of surgery. It is calculated on the basis of a standardized physical examination by the physician. This clinical examination assesses six criteria and differs slightly between the upper and lower limb. For the lower limb, the components are pain, function, emotional acceptance of the treatment outcome, need for walking aids, walking and gait. For all criteria, the estimate is made from bad to very good with parallel awarding of points (0 to 5). There is thus a numerical value for each of the six criteria. These six values are added and divided by the maximum possible number of points (30). The percentage value is obtained by multiplying the calculated point value by 100.

The painDETECT questionnaire (PD-Q) is a quick, simple and reliable screening tool to identify the likelihood of a neuropathic pain component in patients with neuropathic pain. This questionnaire had been prepared by professionals and validated in various languages including Hindi and Marathi. Its sensitivity and specificity is higher than other screening questionnaires for neuropathic pain, including the Douleur Neuropathique 4 (DN4), Leeds Assessment of Neuropathic Symptoms and Signs (LANNS), and the Neuropathic Pain Questionnaire (NPQ) (Freynhagen et al 2006). The PD-Q has been used to identify neuropathic pain in patients with knee osteoarthritis (Ohtori et al 2012) and to identify sensory proﬁles in patients with diabetic neuropathy and postherpetic neuralgia (Baron et al 2009).This questionnaire will be administered tot he patients preoperatively , at 1, 4 and 6 months after surgery.

Details of postoperative chemotherapy and radiation will also be obtained from patient's notes and the electronic medical record. If the patient cannot follow up at the said intervals, the pain scores would be obtained telephonically and the BPI and PD-Q forms in prepaid envelopes would be given to them at discharge which they would have to duly fill in and post them to the given address at the appropriate intervals if they cannot visit the pain clinic. At the 6th month of follow up, they would be requested to visit the pain clinic for an assessment of MSTS score and completing the BPI and PD-Q.

MEASUREMENTS:-

* All demographic, preoperative, intraoperative and postoperative data would be collected by the investigators.
* Demographic data includes case no, age, sex, ASA (American Society of Anesthesiologists) grade.
* Preoperative variables include pain score, preoperative analgesics, duration of use, and the dose.
* Intraoperative variables include duration of surgery, tourniquet time, any nerve or muscle resection and length of bone resected.
* Postoperative variables include median average and worst pain score for the first 3 postoperative days , 1, 4 and 6 months after surgery.
* Analgesics administered postoperatively, dose & dosing intervals, impact on daily functions as obtained from the BPI pre-operatively, 1, 4 and 6 months postoperatively.
* The painDETECT score to identify the neuropathic component of pain if any, preoperatively and at 1, 4 and 6 months after surgery.
* The MSTS score calculated by the physician and obtained from the patient's record at the 6th month after surgery.

STATISTICAL ANALYSIS:- The above mentioned data will be presented as mean (sd), median (range), and frequency (percentage). Categorical data will be analyzed using the Chi-square test or Fisher Exact test (for binary data). Continuous variables will be analyzed using paired t test or Wilcoxon signed rank test as per distribution of data. Repeated measure ANOVA will be used for pain score analysis. Pearson correlation coefficients will be used for association. p-value <0.05 will be considered statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years of age, undergoing TKR
* Literate: able to read and write in at least one of the following languages English, Hindi and Marathi
* Willing to fill forms and post them and/or answer questions on phone

Exclusion Criteria:

* Refusal of consent
* Cognitively impaired
* Revision knee arthroplasty (including cases with wound wash and nail spacer cementing)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for total knee arthroplasty for osteogenic sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
pain severity in the immediate post-operative period following oncologic TKRs | First 3 postoperative days
  Pain scores as per the numerical rating scale

SECONDARY OUTCOMES:
the proportion of patients who continue to have pain at 4 and 6 months post surgery(CPSP) | 4 and 6 months after surgery
  As assessed from the brief pain inventory
• To identify the type of pain (neuropathic component) persisting at 4 and 6 months after TKR | 4 and 6 months from surgery
  Neuropathic component to be identified by using the pain Detect
Impact of the pain on daily function | 4 and 6 months after surgery
  Brief pain inventory and the MSTS score to assess the interference of pain with daily function and how it compares with MSTS at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: APARNA S CHATTERJEE, MD,FCARCSI, Principal Investigator — Professor
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen MP, Buckwalter JA, Miller BJ. Patterns of improvement following oncologic reconstructrion compared to total knee arthroplasty and revision knee arthroplasty. Iowa Orthop J. 2011;31:160-5. PMID 22096436
- [Background] Beswick AD, Wylde V, Gooberman-Hill R. Interventions for the prediction and management of chronic postsurgical pain after total knee replacement: systematic review of randomised controlled trials. BMJ Open. 2015 May 12;5(5):e007387. doi: 10.1136/bmjopen-2014-007387. PMID 25967998
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Ayers DC, Franklin PD, Ploutz-Snyder R, Boisvert CB. Total knee replacement outcome and coexisting physical and emotional illness. Clin Orthop Relat Res. 2005 Nov;440:157-61. doi: 10.1097/01.blo.0000185447.43622.93. PMID 16239800
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Tunn PU, Pomraenke D, Goerling U, Hohenberger P. Functional outcome after endoprosthetic limb-salvage therapy of primary bone tumours--a comparative analysis using the MSTS score, the TESS and the RNL index. Int Orthop. 2008 Oct;32(5):619-25. doi: 10.1007/s00264-007-0388-8. Epub 2007 Aug 15. PMID 17701173
- [Background] Mathieson S, Lin C. painDETECT questionnaire. J Physiother. 2013 Sep;59(3):211. doi: 10.1016/S1836-9553(13)70189-9. No abstract available. PMID 23896340
- [Background] Jain P, Padole D, Bakshi S. Prevalence of acute neuropathic pain after cancer surgery: A prospective study. Indian J Anaesth. 2014 Jan;58(1):36-42. doi: 10.4103/0019-5049.126788. PMID 24700897